CLINICAL TRIAL: NCT05796323
Title: Perceptions and Prevalence of Workplace Violence in Healthcare
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 009.NUR.2022.A
Record Dates: First submitted 2023-02-16; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Violence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Methodist Health System Employees: All MHS employees, clinical and non-clinical.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — The subjects will complete a survey related to workplace violance.

SUMMARY:
Workplace violence includes physical and verbal aggression as well as threatening behavior. All types of workplace violence incidents in health care are often under-reported, especially if there is no lasting physical injury.

DETAILED DESCRIPTION:
Research reveals that healthcare workers are three times more likely to experience workplace violence than any other occupation. The first step toward reducing the occurrence of violence is to understand the perceptions and prevalence of workplace violence.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be employed full-time, part-time, or per diem

Exclusion Criteria:

* Inability to read English will cause a staff member to be excluded from the study, as the survey is written in English.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must be employed full-time, part-time, or per diem (PRN) by the acute care organization (MDMC, MCMC, MMMC, MSMC, MLMC) at the time of study data collection. All staff, both clinical and non-clinical, are eligible to participate. Participants must be able to read English.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-16 (Estimated); Study Completion 2024-03-16 (Estimated)

PRIMARY OUTCOMES:
Level and type of workplace violence | Period of 6 months
  Research Instruments Survey Questionnaire used to measure physical and psychological characteristics of violence at work
Impact on the individual employee/worker | Period of 6 months
  Self-reported consequences in relation to work (e.g., distress/burnout, transfer/quits, absenteeism, financial situation, career path)

SECONDARY OUTCOMES:
Research Instruments Survey Questionnaire | Period of 6 months
  Survey Monkey will be used to measured Frequency of reported incidents concerning the different forms of violence at work
Self-reported impact of violence on quality of care for patients | Period of 6 months
  Impact on the organization (e.g., cost data, lost work days, staff fluctuation, staff shortage)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sweatt, MSN, RN-BC, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No